CLINICAL TRIAL: NCT07102446
Title: Evaluation of an Opioid Stewardship Program in Non-Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Korea Hospital Pharmaceutical Education & Research Center (Unknown); Korea University (Other)
Responsible Party: Principal Investigator, Lee, So Hyun, Chief of Pharmacy Department, Korea University Guro Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025GR0258
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Pain; Chronic Pain; Opioid Analgesia; Opioid Use
Keywords: Pharmacist; Pain Management; Opioid Stewardship; Non-Cancer Pain
MeSH Terms: conditions — Pain; Chronic Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opioid Stewardship Program Intervention Group (Experimental): Participants in this arm are adult outpatients with chronic non-cancer pain who receive a pharmacist-led Opioid Stewardship Program (OSP) for their chronic opioid use.
  Interventions: Other: Opioid Stewardship Program

INTERVENTIONS:
Other: Opioid Stewardship Program — The Opioid Stewardship Program (OSP) includes pain and functional assessments, opioid prescription review and coordination, patient education, and counseling provided by trained pharmacists.

SUMMARY:
The objective of this prospective, non-randomized clinical trial is to evaluate the effectiveness of a pharmacist-led Opioid Stewardship Program (OSP) in outpatient adults with chronic non-cancer pain. This study compared OSP implementation with a historical control to determine whether it reduces the incidence of high-risk opioid prescribing and improves patients' awareness, knowledge, and attitudes about opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients at the Department of Anesthesiology and Pain Medicine or the Department of Physical Medicine & Rehabilitation of the study site who received a prescription for opioid analgesics (oral, transdermal, sublingual, or buccal formulations containing oxycodone, fentanyl, tapentadol, hydrocodone, or morphine) due to chronic non-cancer pain during the study evaluation period (from IRB approval date to September 30, 2025)
* Adults aged ≥19 years and <80 years
* Patients who voluntarily signed a written informed consent form after receiving a full explanation of the study and understanding its purpose

Exclusion Criteria:

* Patients with active cancer
* Patients diagnosed with sickle cell disease
* Patients diagnosed with a life-limiting illness eligible for hospice or palliative care as defined in Article 2 of the 'ACT ON HOSPICE AND PALLIATIVE CARE AND DECISIONS ON LIFE-SUSTAINING TREATMENT FOR PATIENTS AT THE END OF LIFE'
* Pregnant patients
* Patients who were prescribed opioid analgesics within the past month for postoperative pain management
* Patients who were prescribed opioid analgesics within the past month for newly developed pain
* Patients with communication difficulties
* Patients who were prescribed buprenorphine for the treatment of opioid use disorder
* Patients who are deemed inappropriate for study participation at the discretion of the investigator

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of potentially high-risk opioid prescriptions | At each outpatient visit during the study evaluation period (up to 4 months per participant)
  This outcome measures the proportion of potentially high-risk opioid prescriptions based on predefined criteria:
  * Prescription (Rx) of ER/SR opioids to patients with no prior opioid use
  * Rx of certain ER/SR opioid dosages to patients who are not opioid-tolerant
  * Rx of sublingual/buccal fentanyl
  * Rx exceeding 50 MME/day
  * Rx exceeding 10 MME/dose or 30 MME/day to patients with no prior opioid use
  * Rx with no dose adjustments for the elderly or renally impaired with no prior opioid use
  * ER/SR opioid conversions outside 50-75% of the prior MME/day
  * Rx of oral ER/SR opioids more than twice daily
  * Rx of transdermal fentanyl at intervals less than 72 hours
  * Rx exceeding 30 days supply
  * Rx without a pain assessment in the past 3 months in long-term opioid users
  * No opioid dose adjustment in the last 3 Rx despite additional pain interventions and improved pain in long-term users
  * No opioid dose adjustment in the last 3 Rx despite the lack of pain improvement in long-term users

SECONDARY OUTCOMES:
Average daily morphine milligram equivalent (MME) | At each outpatient visit during the study evaluation period (up to 4 months per participant)
  This outcome assesses the clinical effect of the intervention by calculating the average daily MME for each opioid prescription during the study evaluation period.
Change in opioid knowledge scores after education sessions compared to baseline | At each outpatient visit during the study evaluation period (up to 4 months per participant)
  This outcome evaluates patient understanding of opioid use. Knowledge scores are measured at baseline (before the first education session) and after each of the education sessions using a validated questionnaire.
Change in opioid attitude scores after education sessions compared to baseline | At each outpatient visit during the study evaluation period (up to 4 months per participant)
  This outcome assesses patient attitudes toward opioid use, including concerns about addiction, side effects, and trust in physicians. Attitude scores are measured at baseline and after each of the education sessions using a modified K-PMAQ-14 (Korean version of pain medication attitude questionnaire-14) survey.

CONTACTS AND LOCATIONS:
Overall Officials: So Hyun Lee, MS, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The decision not to share individual participant data (IPD) is based on the possibility that the research data may contain personally identifiable information. Informed consent was not obtained from participants for the sharing of their individual data with third parties.